CLINICAL TRIAL: NCT07220109
Title: A Phase 3, Randomized, Controlled, Observer Blind, Immuno-bridging Study to Evaluate Immunogenicity, Reactogenicity, Safety of a Single Dose of GSK's RSVPreF3 OA Investigational Vaccine in Chinese Adults 18-59 Years of Age at Increased Risk of Respiratory Syncytial Virus Disease
Brief Title: A Study on the Immune Response and Safety of Vaccine Against Respiratory Syncytial Virus Given to Chinese Adults 18 to 59 Years of Age at Increased Risk of Respiratory Syncytial Virus Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 223372
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus (RSV); Immunogenicity; Safety; Reactogenicity; Older adults at increased risk (OA AIR)
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind study: participants the site and sponsor personnel involved in the clinical evaluation of the participants are blinded while the treatment is administered by unblinded study personnel who will not participate in data collection evaluation or review of any study endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSV AIR group (Experimental): Participants at increased risk (AIR) of RSV disease will receive a single dose of investigational RSVPreF3 OA investigational vaccine on Visit 1 (Day 1).
  Interventions: Biological: RSVPreF3 OA vaccine
- Placebo AIR group (Placebo Comparator): Participants AIR of RSV disease will receive a single dose of Placebo on Visit 1 (Day 1).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSVPreF3 OA vaccine — 1 dose of RSVPreF3 OA investigational vaccine administered intramuscularly in the deltoid region of the non-dominant arm.
  Arms: RSV AIR group
Biological: Placebo — 1 dose of saline solution administered intramuscularly in the deltoid region of the non-dominant arm.
  Arms: Placebo AIR group

SUMMARY:
The study will evaluate the immune response of the RSVPreF3 OA investigational vaccine in Chinese adults 18 to 59 years of age (YOA) who are at increased risk of respiratory syncytial virus (RSV) disease, in comparison with the immune response generated in older adults 60 YOA and above from the 219815 (RSV OA=ADJ-021; NCT06551181) study following a single dose of the RSVPreF3 OA vaccine. In addition, the safety and reactogenicity of the vaccine will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed informed consent obtained from the participant (participant must be able to understand the informed consent) prior to performance of any study-specific procedure.
* A male or female participant 18-59 YOA at the time of the study intervention administration.
* Participants should be diagnosed with at least 1 of the following medical conditions if considered medically stable* by the investigator:

  * A stable condition is defined as a disease not requiring significant change (based on the investigator's opinion) in therapy or worsening during the 3 months before enrollment.

    -Chronic cardiopulmonary disease resulting in activity restricting symptoms or use of long-term medication: oChronic obstructive pulmonary disease (COPD)
* Global Initiative for Chronic Obstructive Lung Disease (GOLD) Grade 2-4 oAsthma
* Patient on Maintenance and Reliever Therapy (MART) OR with at least one rescue treatment per week (excluding exercise asthma) oCystic fibrosis oOther chronic respiratory diseases: lung fibrosis, restrictive lung disease, interstitial lung disease, emphysema or bronchiectasis oChronic heart failure:
* A minimum of class II symptoms according to New York Heart Association classification of heart failure oPre-existing CAD (CAD not otherwise specified)
* Physician diagnosis of CAD based on electrocardiogram, exercise stress test, nuclear stress test, cardiac computed tomography scan or cardiac angiogram (more than the presence of hypercholesterolemia) oCardiac arrhythmia
* Patient diagnosed with a cardiac arrythmia that require medical support either pharmacologically or with a medical device -Diabetes mellitus: types 1 or 2 with active treatment for the past 6 months

  -Other diseases at increased risk for RSV disease oChronic kidney disease
* G2-G3 disease (Glomerular Filtration Rate between 30 and 90 mL/min/1.73 m2) oChronic moderate to severe liver disease
* Female participants of non-childbearing potential may be enrolled in the study. Non childbearing potential is defined as premenarche, hysterectomy, bilateral oophorectomy, bilateral salpingectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception from 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study prior to intervention administration, and
  * has agreed to continue adequate contraception for at least 1 month after completion of the study intervention administration.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention
* Unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent or uncontrolled neurological disorders or seizures. Participants with medically controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol. Study participants may decide to assign a caregiver to help them complete the study procedures.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

•Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study intervention during the period beginning 30 days before the dose of study intervention (Day -29 to Day 1), or planned use during the study period (up to Contact, Month 6).

* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after the dose of study intervention administration, with the exception of inactivated, subunit and split influenza vaccines or COVID-19 vaccines which can be administered up to 14 days before or from 14 days after the study intervention administration.
* Previous vaccination with any RSV vaccine, including investigational RSV vaccines.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or administration of long-acting immune-modifying treatments or planned administration at any time up to the EOS.

  * Up to 3 months prior to the study intervention administration:

oFor corticosteroids, this will mean prednisone >=20 mg/day, or equivalent. Inhaled, topical and intra-articular steroids are allowed oAdministration of immunoglobulins and/or any blood products or plasma derivatives -Up to 6 months prior to study intervention administration: long-acting immune-modifying drugs including among others immunotherapy, monoclonal antibodies, antitumoral medication.

Prior/Concurrent clinical study experience

•Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or invasive medical device).

Other exclusion criteria

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Bedridden participants.
* Planned move during the study conduct that prohibits participation until study end.
* Participation of any study personnel or their immediate dependents, family, or household members.
* Pregnant or lactating female participant.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 1 month after study intervention administration.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
RSV-A neutralizing titers expressed as group Geometric Mean Titers (GMTs) | At Day 31 (i.e., 1 month after RSVPreF3 OA investigational vaccine administration)
  The serum neutralizing titers are expressed in Estimated Dilution (ED60). The group GMT ratio will be evaluated for RSV-OA overseas group (from RSV OA-ADJ-021 study) over RSV AIR (from the current study).
RSV-A neutralizing titers expressed as group Seroresponse rate (SRR) | At Day 31 (i.e., 1 month after RSVPreF3 OA investigational vaccine administration)
  The SRR is defined as the proportion of participants having a 4-fold increase in neutralizing titers. The group SRR difference will be evaluated for RSV-OA overseas group (from RSV OA-ADJ-021 study) minus RSV AIR (from the current study).
RSV-B neutralizing titers expressed as group GMTs | At Day 31 (i.e., 1 month after RSVPreF3 OA investigational vaccine administration)
  The serum neutralizing titers are expressed in ED60. The group GMT ratio will be evaluated for RSV-OA overseas group (from RSV OA-ADJ-021 study) over RSV AIR (from the current study).
RSV-B neutralizing titers expressed as group SRR | At Day 31 (i.e., 1 month after RSVPreF3 OA investigational vaccine administration)
  The group SRR difference will be evaluated for RSV-OA overseas group (from RSV OA-ADJ-021 study) minus RSV AIR (from the current study).

SECONDARY OUTCOMES:
RSV-A and RSV-B neutralizing titers expressed as group GMTs | At Day 31 and at Month 6 (i.e., 1 month and 6 months after RSVPreF3 OA investigational vaccine administration)
  The serum neutralizing titers are expressed in ED60. The group GMT ratio will be evaluated for RSV-OA Chinese group (from RSV OA-ADJ-021 study) over RSV AIR (from the current study).
RSV-A and RSV-B neutralizing titers expressed as group SRR | At Day 31 and at Month 6 (i.e., 1 month and 6 months after RSVPreF3 OA investigational vaccine administration)
  The group SRR difference will be evaluated for RSV-OA Chinese group (from RSV OA-ADJ-021 study) minus RSV AIR (from the current study).
Number of participants with RT-PCR-confirmed RSV A and/or B-associated acute respiratory illness (ARI) and lower respiratory tract disease (LRTD), assessed for all groups of the current study | Day 1 to Month 6 of the current study
  An ARI is defined as the presence of at least 2 respiratory symptoms/signs for at least 24 hours; or at least 1 respiratory symptom/sign and 1 systemic symptom/sign for at least 24 hours. An RT-PCR-confirmed RSV-ARI is an event meeting the case definition of ARI with at least one RSV-positive swab detected by RT-PCR. A LRTD is defined as the presence of at least 2 lower respiratory symptoms/signs for at least 24 hours including at least 1 lower respiratory sign; or at least 3 lower respiratory symptoms for at least 24 hours. An RT-PCR-confirmed RSV-LRTD is an event meeting the case definition of LRTD with at least one RSV-positive swab detected by RT-PCR.
Duration of RT-PCR-confirmed RSV A and/or B-associated ARI and LRTD episodes, assessed for all the groups of the current study | Day 1 to Month 6 of the current study
Number of participants reporting symptoms/signs of RT-PCR-confirmed RSV A and/or B-associated ARI and LRTD, assessed for all the groups of the current study | Day 1 to Month 6 of the current study
Number of participants with RT-PCR-confirmed RSV A and/or B-associated ARI and LRTD by severity, assessed for all the groups of the current study | Day 1 to Month 6 of the current study
Number of participants with RT-PCR-confirmed RSV A and/or B-associated ARI and LRTD by frailty status, assessed for all the groups of the current study | Day 1 to Month 6 of the current study
Number of participants with each solicited administration site event assessed for all the groups of the current study | Day 1 to Day 7 of the current study
  Solicited administration site event are pain, erythema and swelling.
Number of participants with each solicited systemic event assessed for all the groups of the current study | Day 1 to Day 7 of the current study
  Solicited systemic events are fever, myalgia (muscle pain), arthralgia (joint pain), headache and fatigue (tiredness). Fever is defined as a temperature of more than or equal to (>=) 38.0 degrees Celsius (°C).
Number of participants with unsolicited adverse events (AEs) assessed for all the groups of the current study | Day 1 to Day 30 of the current study
  An unsolicited AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Number of participants with serious adverse events (SAEs) assessed for all the groups of the current study | Day 1 up to study end (Month 6) of the current study
  An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, abnormal pregnancy outcomes, is a suspected transmission of any infectious agent via an authorized medicinal product. or any other situation considered as such by the investigator.
Number of participants with potential immune-mediated disease (pIMDs) assessed for all the groups of the current study | Day 1 up to study end (Month 6) of the current study
  PIMDs are a subset of adverse events of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - GSK Investigational Site, Xiangtan, Hunan
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf